CLINICAL TRIAL: NCT01484249
Title: Carotid Filtration During Endovascular Aortic Valve Implantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Claret Medical (Industry)
Collaborators: Meditrial Europe Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CMP 001b
Record Dates: First submitted 2011-11-24; First posted 2011-12-02 (Estimated); Last update posted 2011-12-05 (Estimated); Status verified 2011-12

CONDITIONS: Heart Diseases
Keywords: embolic; filters; brachiocephalic; neurovasculature; debris
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: CE Pro System — The CE Pro System consists of a delivery catheter with an integrated proximal filter intended to be deployed in the brachiocephalic artery. In addition, the device has an articulating distal tip and a through lumen to allow a commercial intravascular filter to be back-loaded into the CE Pro System and be deployed into and retrieved from the left carotid artery.
  Other Names: Gen 2.0; Gen 2.1; Gen 2.2

SUMMARY:
This study was designed as a First In Man (FIM) trial to evaluate the feasibility and technical capability of the Claret CE Pro System in delivering two embolic filters to the brachiocephalic artery and the left common carotid artery during a Transcatheter aortic valve implantation (TAVI) procedure in order to protect the neurovasculature from debris liberated during the procedure.

DETAILED DESCRIPTION:
Transcatheter aortic valve implantation (TAVI) is a recently developed procedure whereby a prosthetic aortic valve is implanted percutaneously, and the procedure has demonstrated promising results in high risk surgical populations.

TAVI currently requires the use of large bore (18-26F) catheter delivery systems that are often difficult to deliver to over the aortic arch to the aortic annulus. Available data indicate that TAVI is associated with a 4-12% procedural stroke rate and approximately 10% procedural mortality. It has been suggested that these strokes are most likely caused by the liberation of embolic debris either when the TAVI delivery catheter is advanced over the aortic arch or during the actual valve deployment. Given this situation, the availability of devices able to protect both hemispheres of the brain from potentially embolic debris during the TAVI procedure is an emerging clinical need.

Claret Medical has developed a technology to provide protection to the neurovascular system during TAVI and other valve repair procedures.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be scheduled to undergo an endovascular aortic valve prosthesis implant procedure with the femoral artery as the intended access site for the valve delivery system.
* Female subjects of child bearing potential must have a negative pregnancy test within 48 hours prior to the study procedure.
* Subject's left carotid artery and innominate artery diameters must be compatible with the Claret CE Pro System sizes available for the procedure (refer to package labeling for appropriate sizing information).
* Subject must have been informed of the nature of the study, agree to its provisions, and provide written informed consent.

Exclusion Criteria:

* Subject requires an emergent procedure.
* Subject has carotid artery stenosis >70% in either carotid artery.
* Subject innominate or left carotid artery reveals significant stenosis, ectasia, dissection or aneurysm at the ostium or within 3 cm of the ostium.
* Subject has allergy to materials from which the device is constructed (Nitinol, fluorinated ethylene-propylene, polyamide, polyimide, platinum, iridium, stainless steel, cyanoacrylate adhesives, polycarbonate, polyethylene, polyester, polyurethane, PTFE [poly-tetrafluoroethylene], polydimethylsiloxane [lubricant coating], silicone, polyetheretherketone, tin-silver [solder] or acrylated urethane adhesives)
* Subject has a history of bleeding diatheses or coagulopathy or will refuse blood transfusion in cases of emergency.
* Subject has renal insufficiency, defined as a creatinine level > 2.5 mg/dl at the time of treatment, unless subject is on chronic hemodialysis.
* Subject has hyperthyroidism.
* Subject suffered recent (within the past 3 months) stroke with permanent deficit.
* Subject suffered recent (within the past 6 months) significant gastrointestinal (GI) bleed.
* Subject is involved in another clinical study or has other medical illnesses that may cause the subject to be non-compliant with the protocol or confound the data interpretation.
* Subject history of intolerance, allergic reaction or contraindication to any of the study medications, including heparin, aspirin, Clopidogrel, or a sensitivity to contrast media or anesthesia which cannot be adequately pre-treated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2010-02; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Primary endpoint is technical success of the CE Pro System to deliver, retrieve proximal & distal filters during an endovascular procedure such as Transcatheter aortic valve implantation (TAVI). | From the CE Pro System Insertion Start Time to Final Retrieval Stop Time
  Technical success defined as, successful delivery & retrieval of the proximal & distal filters.
  The following Operator feedback was collected & used to evaluate the primary endpoint.
  Operators are asked to record, the indwelling time for the CE Pro System was used. Calculated as duration from the CE Pro System Insertion Start Time to Final Retrieval Stop Time.
  Operators are asked to rate the CE Pro Systems performance based on a scale of 1 to 5, with 5 being the highest rating.

SECONDARY OUTCOMES:
Transient Ischemia Attack (TIA) Rates | 30 day follow up
  The secondary endpoints for this trial are safety endpoints and are presented as adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Eberhard Grube, MD, Ph D, Principal Investigator — Professor of Medicine, Medizinishce Klinik und Poliklinik II, Universitätsklinikum Bonn